CLINICAL TRIAL: NCT02997605
Title: Comparison of Two Strategies of Glucocorticoid Withdrawal in Rheumatoid Arthritis Patients in Low Disease Activity or Remission.
Brief Title: Comparison of Two Strategies of Glucocorticoid Withdrawal in Rheumatoid Arthritis Patients
Acronym: STAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RC31/15/7824; 2016-001618-18 (EudraCT Number); PHRC (Other Grant/Funding Number: French Ministry of Health)
Record Dates: First submitted 2016-12-15; First posted 2016-12-20 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2022-02

CONDITIONS: RheumatoId Arthritis
Keywords: low disease activity; remission
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Glucocorticoids; Prednisone; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucocorticoid (GC) tapering (Active Comparator): "GC tapering group": patients will be asked to taper prednisone taken every morning at 8.00 AM by decreasing the daily dose by 1 mg every month as soon as they are in remission or Low Disease Activity (LDA). In addition they will receive a placebo of 20 mg/day of hydrocortisone (10 mg at 8.00 AM, 10 mg at 12.00 AM) for 3 months then 10 mg/day (at 8.00 AM) of hydrocortisone placebo for 3 months before discontinuing the hydrocortisone placebo.
  Interventions: Drug: GlucoCorticoid
- Hydrocortisone replacer (Active Comparator): "Hydrocortisone replacer group": patients will replace prednisone with 20 mg of hydrocortisone on a daily basis (10 mg at 8.00 AM, 10 mg at 12.00 AM) for 3 months then 10 mg daily (at 8.00 AM) for 3 months then stop as soon as they are in remission or LDA, as well as a prednisone placebo (at 8.00 AM) with a schedule to taper the prednisone placebo by 1mg/day every month until discontinuation.
  Interventions: Drug: GlucoCorticoid

INTERVENTIONS:
Drug: GlucoCorticoid — After inclusion in the study, the first part is an open follow-up period where all patients will receive 5 mg of prednisone daily for one month. After one month, if patients still have a DAS28 ≤3.2, they will be randomized into two arms: Group 1: "GC tapering group" / Group 2: "Hydrocortisone replacement group".
  After randomisation, there are four scheduled visits: M4, M7, M9 and M12. Patients withdrawing from GC therapy will be instructed, that if they start feeling unwell during or after the GC tapering protocol they should not taper the steroid dose any further, but contact the centre responsible for the protocol. If GC induced adrenal insufficiency is confirmed or strongly suspected, GC replacement will be secured using hydrocortisone.
  Other Names: Prednisone, Hydrocortisone

SUMMARY:
The purpose of this study is to compare the proportion of patients who could withdraw from prednisone and hydrocortisone one year after a progressive decrease of GC (GC tapering) or a hydrocortisone replacement therapy in rheumatoid arthritis in remission or low disease activity.

DETAILED DESCRIPTION:
French multicenter double-blind controlled parallel-group randomized clinical trial Phase IV assessing whether a hydrocortisone replacement therapy could increase the success rate of GC withdrawal at one year, in patients with Rheumatoid Arthritis in low disease activity or remission, in comparison to progressive decrease of GC (GC tapering).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old.
* Fulfilling the 2010 American College of Rheumatology (ACR)/EULAR criteria for RA.
* Treated with a stable dose of Synthetic Disease Modifying Anti-Rheumatic Drugs (sDMARD) or Biological Disease Modifying Anti-Rheumatic Drug (bDMARD) for at least 3 months.
* Who have been treated with prednisone or prednisolone for at least 6 months.
* With a stable dose of prednisone or prednisolone of 5mg/day for at least 3 months.
* With a DAS28 ≤3.2 for at least 3 months.
* Patients with health insurance
* Patients who have signed a written informed consent form.

Exclusion Criteria:

* Any chronic condition that would need long term corticoid use (e.g. chronic lung diseases).
* Evidence of a flare within the last 3 months.
* Evidence of an allergy or intolerance to hydrocortisone or prednisone.
* Chronic idiopathic, or autoimmune clinical adrenal insufficiency.
* GC joint injections within the last 3 months or scheduled in the next 3 months.
* Any GC intake expected more than >5mg/day within the next 12 months.
* Association with sultopride and with live vaccines
* Significant trauma or major surgery within the 3 months prior to the baseline visit.
* Scheduled surgery in the next 12 months.
* Fibromyalgia.
* Foreseeable poor compliance with the strategy.
* Patient with any condition that would prevent participation in the study and completion of the study procedures, including language limitation.
* Alcohol and/or drug misuse as determined by the investigator.
* Pregnancy or breastfeeding.
* Patient is not willing to sign the informed consent.
* Juridical Protection
* DAS28>3.2 after one month of a stable dose of prednisone 5 mg/day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
proportion of patients who could withdraw from prednisone and hydrocortisone at one year | one year after a progressive decrease of Glucocorticoids or hydrocortisone replacement
  To compare a prednisone tapering strategy to a hydrocortisone replacement strategy on the success rate of prednisone and hydrocortisone withdrawal at one year in Rheumatoid Arthritis patients in low disease activity or remission.

SECONDARY OUTCOMES:
proportion of patients who could withdraw from prednisone | one year after a progressive decrease of Glucocorticoids or hydrocortisone replacement
  To compare the proportion of patients who could withdraw from prednisone whatever the additional hydrocortisone associated treatment.
proportion of patients with acute adrenal insufficiency | one year
  To compare the proportion of patients with acute adrenal insufficiency at one year between the two groups.
proportion of patients with biological adrenal insufficiency | one year
  To compare the proportion of patients with biological adrenal insufficiency at one year between the two groups.
proportion of patients needing extra prednisone to control flares | one year
  To compare the proportion of patients needing extra prednisone to control flares
proportion of patients who have at least one flare confirmed by the investigator during the protocol. | one year
  To compare the proportion of patients who have at least one flare confirmed by the investigator during the protocol.
area under the curve of means of the FLARE (Flare Assessment in Rheumatoid Arthritis) | one year
  To compare the area under the curve of the means of the FLARE (Flare Assessment in Rheumatoid Arthritis) at one year with a self-assessment questionnaire.
proportion of patients in DAS28 remission and in DAS28 low disease activity | 7 and 12 months
  To compare the proportion of patients in DAS28 remission and in DAS28 low disease activity at 7 and 12 months between the groups.
medians of Health Assessment Questionnaire (HAQ) | 4, 7 months and 1 year
  To compare the medians of HAQ at 4, 7 months and one year between the groups.
medians of Rheumatoid Arthritis Impact of Disease (RAID) | 4, 7 months and 1 year
  To compare the medians of RAID at 4, 7 months and one year between the groups.
medians of EuroQol 5-dimensional Descriptive system (EQ-5D) | 4, 7 months and 1 year
  To compare the medians of EQ-5D at 4, 7 months and one year between the groups.
medians of Functional Assessment of Chronic Illness Therapy - Fatigue Scale FACIT-F) | 4, 7 months and 1 year
  To compare the medians of FACIT-F at 4, 7 months and one year between the groups.
proportion of patients with Serious Adverse events | 1 year
  To compare the proportion of patients with Serious Adverse events at one year between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Adeline RUYSSEN-WITRAND, MD, PhD, Study Chair — University Hospital of Toulouse, Rheumatology Center; Arnaud CONSTANTIN, MD, PhD, Study Chair — University Hospital of Toulouse, Rheumatology Center
Locations (17):
- France (17):
  - Bordeaux University Hospital, Bordeaux
  - Brest University Hospital, Brest
  - Jean Rougier Hospital, Cahors
  - Clermont-Ferrand Hospital, Clermont-Ferrand
  - Bicêtre Hospital, Le Kremlin-Bicêtre
  - Lille Hospital, Lille
  - Limoges Hospital, Limoges
  - Montpellier Hospital, Montpellier
  - Pasteur Hospital, Nice
  - Orléans Hospital, Orléans
  - Bichat Hospital, Paris
  - Cochin Hospital, Paris
  - La Pitié-Salpétrière, Paris
  - Lyon Sud Hopsital, Pierre-Bénite
  - Saint-Etienne Hospital, Saint-Etienne
  - Strasbourg Hospital, Strasbourg
  - Hospital Pierre-Paul Riquet, Toujouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ruyssen-Witrand A, Brusq C, Masson M, Bongard V, Salliot C, Poiroux L, Nguyen M, Roux CH, Richez C, Saraux A, Vergne-Salle P, Morel J, Flipo RM, Piperno M, Gottenberg JE, Marotte H, Soubrier M, Gossec L, Dieude P, Lassoued S, Zabraniecki L, Couture G, Boyer JF, Jamard B, Degboe Y, Constantin A. Comparison of two strategies of glucocorticoid withdrawal in patients with rheumatoid arthritis in low disease activity (STAR): a randomised, placebo- controlled, double-blind trial. Ann Rheum Dis. 2025 Jan;84(1):49-59. doi: 10.1136/ard-2024-226620. Epub 2025 Jan 2. PMID 39874233